CLINICAL TRIAL: NCT04346056
Title: Retrospective Study From November 2019 -Febrauary 2020 on Severe Respiratory Illness to Access the Presence or Absence of COVID-19 in Patients Samples by Real-time PcR
Brief Title: Retrospective Study on Severe Respiratory Illness to Access the Presence of COVID-19
Acronym: Explore
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Hassan Agwa, Consultant of Clinical pathology & Molecular genomics, Ain Shams University
Other Study IDs: FMASU P17a/ 2020
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Disease (COVID-19); COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Oropharyngeal and nasopharyngeal swabs for hospitalized SARI patients who meet the WHO standard SARI case definition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective study from November 2019 -Febrauary 2020 on severe respiratory illness to access the presence or absence of COVID-19 in patients samples by real-time PcR

DETAILED DESCRIPTION:
A- Methodology adopted in the retrospective study:

Sample Size Determination:

500 case presented from November 2019- February 2020 will be included in explore study from Ain shams university Hospitals

Collection of Samples:

Oropharyngeal and nasopharyngeal swabs (NP) for hospitalized SARI patients:

Clinicians in the internal medicine, chest, and pediatric hospitals will be responsible for obtaining oropharyngeal and nasopharyngeal swabs for laboratory testing from all hospitalized patients who meet the WHO standard SARI case definition.

Oropharyngeal swabbing:

A dry sterile tip flocked with nylon fiber swab applicator should be used to swab the posterior pharynx. The swab should be placed in a 15 ML centrifuge tube labeled with the patient unique ID and containing 2mL viral transport media (VTM). The applicator stick is then cut off.

Nasopharyngeal swabbing:

A flexible, sterile tip flocked with nylon fiber swab applicator is inserted into the nostril and back to the nasopharynx and left in place for a few seconds. It is then slowly withdrawn with a rotating motion. For SARI patients, the swab is put into the same centrifuge tube as the oropharyngeal swab labeled with the patient's unique ID and the shaft is cut. The 15 ml tube containing the swab/s should be carefully transported to the hospital laboratory as soon as possible in cold chain.

Sample processing:

The received swabs inside the 15 ml tube should be agitated vigorously for 10 seconds using a vortex mixer to free cells from the swab tip, and then both swabs should be removed from the tube and discarded using a forceps. The VTM should be split into 2 pre-labeled, sterile cryovials with the correct patient ID. One cryovial should be immediately placed in a freezer (-70°C), while the other cryovial will be used the molecular testing by real time PCR at MASRI-molecular laboratory.

Samples will be tested by real time multiplex PCR using FTD- respiratory 33 kit for the presence of a wide panel of respiratory pathogens that include: influenza A and subtypes influenza A Pdm(H1N1) and seasonal H3, influenza B, influenza C, parainfluenza viruses 1, 2, 3 and 4; coronaviruses NL63, 229E, OC43 and HKU1; human metapneumoviruses A and B; rhinovirus; respiratory syncytial viruses A and B ; adenovirus; enterovirus; parechovirus; Boca virus; Pneumocystis jirovecii; Mycoplasma pneumoniae; Chlamydia pneumoniae; Streptococcus pneumoniae; Haemophilus influenza type B (HIB assay also detects Haemophilus parahaemolyticus which is associated with pharyngitis); Staphylococcus aureus; Moraxella catarrhalis; Bordetella spp. (except Bordetella parapertussis), Klebsiella pneumoniae; Legionella species and Salmonella species. Cases suspected with MERS-CoV or HPAI H5N1 according to their history of contact with birds or camels or with reference to the WHO suspected cases of MERS-CoV or avian influenza will be tested using the CDC protocol.

Sample storage:

The second aliquot of the samples will be stored in freezers (-70°C) at MASRI MOLECULAR laboratory for External Quality Assurance (EQA) by on site testing through random selection of samples with different results and retest them by other NAMRU-3 laboratory expertise in MASRI molecular labs; the samples can also be used for further testing by NGS or virus isolation in MASRI molecular laboratories.

Sample Transfer:

All samples will be kept in Faculty of Medicine Ain Shams Research Institute- Molecular Unit laboratories and will not be transferred to other laboratories.

B- Explore study testing for COVID-19 using ready to use RT-real time test assays - VIRAL RNA ISOLATION: Using commercially available kits supplied by thermofisher or other recommended companies. Work will be done in Biosafety level 2 cabinets under complete sterile conditions. -

COVID-19 DETECTION:

Using real-time reverse transcription polymerase chain reaction RT-PCR the test can be done on respiratory samples obtained by various methods, including nasopharyngeal swab or sputum sample. Results are generally available within a few hours. Molecular methods leverage polymerase chain reaction (PCR) along with nucleic acid tests, and other advanced analytical techniques, to detect the genetic material of the virus using real-time reverse transcription polymerase chain reaction for diagnostic purposes. Commercially available kits supplied by hvd, thermofisher and others.

C- Genome sequencing (NGS) for possible positive covid-19 samples Ion Torrent targeted next-generation sequencing (NGS) enables a streamlined research workflow for complete genome sequencing and epidemiological studies of SARS-CoV-2 (the coronavirus responsible for COVID-19). Through the use of a set of highly specific, universal coronavirus primers in combination with a high-fidelity master mix, all genomic segments are amplified and the DNA amplicons are sequenced on any Ion Torrent system to deliver highly accurate coronavirus typing in under a day. The Ion ArnpliSeq SARS-CoV-2 Research Panel consists of 2 pools with arnplicons ranging from 125275 bp iri length for complete viral genome sequencing

ELIGIBILITY:
Inclusion Criteria:

* 500 case presented from November 2019-February 2020 will be included in explore study from Ain shams university Hospitals

Exclusion Criteria:

* Inadequate samples

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hospitalized patients who meet the WHO standard SARI case definition
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Exploring the presence of COVID-19 | 9 months
  Exploring the presence of COVID-19 in very well preserved oropharyngeal samples since November 2019

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hassan, Principal Investigator — Ain Shams University
Locations (2):
- Egypt (2):
  - Faculty of Medicine Ain Shams University, Cairo, Non-US
  - Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US

IPD SHARING:
Plan to Share IPD: No